CLINICAL TRIAL: NCT04545931
Title: Posterior Tibial Nerve Stimulation Vs Desmopressin In Children With Primary Monosymptomatic Nocturnal Enuresis
Acronym: PTNS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud S Amar, MD, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M5_64_2020
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Primary Monosymptomatic Nocturnal Enuresis
Keywords: Nocturnal enuresis, PTNS, effect
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: patient will be allocated to either arms of the study using concealed random allocation method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Posterior tibial nerve stimulation (Experimental): First arm will undergo posterior tibial nerve stimulation ( one session per week for 12 weeks )
  Interventions: Device: Posterior tibial nerve stimulation
- Desmopressin (Experimental): Second arm will receive medical treatment (desmopressin 0.2 mg . single evening dose ) for 12 weeks
  Interventions: Drug: Desmopressin Acetate

INTERVENTIONS:
Device: Posterior tibial nerve stimulation — 34-gauge stainless steel needle is inserted about three finger breadths cephalad to the medial malleolus. In children, previous administration of a topical anesthetic agent (e.g. lidocaine) can help to reduce pain and fear associated with needle insertion. The goal is to place the tip of the needle close to the PTN without actually touching it. The negative electrode is placed on the same leg near the arch of the foot. The needle and the electrode are connected to a low voltage (9 V) stimulator
  Other Names: Urgent PC
  Arms: Posterior tibial nerve stimulation
Drug: Desmopressin Acetate — 0.2 mg, single evening dose ) for 12 weeks, tapering to half of the dose daily for two weeks before discontinuation
  Arms: Desmopressin

SUMMARY:
Nocturnal enuresis is a worldwide health problem frequently encountered in childhood . It affects 18 % of younger school- age children in Egypt. It is the most frequent (85%) type of enuresis in children (Eberdt-Gołabek et al, 2013), . Nocturnal enuresis includes monosymptomatic nocturnal enuresis with no day time urinary symptoms and non monosymptomatic nocturnal enuresis that accompanied by day time urinary symptoms . It can cause severe psychological and social distress to children and their parents . The currently recommended treatment such as alarms , antidiuretic hormone and anticholenergics are not effective in all children with significant relapse rate . Although it's mechanism of action is not fully elucidated , posterior tibial nerve stimulation is safe and acceptable, with evidence of potential clinical effect for both bladder and bowel dysfunction (Bellette et al, 2009). This study will investigate the effect of posterior tibial nerve stimulation on primary monosymptomatic nocturnal enuresis in children.

DETAILED DESCRIPTION:
Nocturnal enuresis is a worldwide health problem frequently encountered in childhood. 85% of cases of nocturnal enuresis are primary mono-symptomatic nocturnal enuresis that can cause substantial psychological impact on children and their families. The currently recommended treatment for NE are not effective in all children with high relapse rate. Posterior tibial nerve stimulation was introduced with early promising results as neuro-modulative therapy for both bladder and bowel dysfunction, although it's mechanism of action is not fully understood.

This study aims to assess the efficacy and role of posterior tibial nerve stimulation versus Desmopressin in primary mono-symptomatic nocturnal enuresis.

80 patients with PMNE were included, over a period of 6 months, at Urology department of Abou ElRish Children's Hospitals, Cairo University. The patients were divided into 2 groups, first group underwent posterior tibial nerve stimulation ( one session per week for 12 weeks ) and the other group of patients received medical treatment (Desmopressin 0.2 mg, single evening dose) for 12 weeks. Both groups are constructed to be adherent to behavioral therapy. The two groups were statistically evaluated regarding the frequency of nocturnal enuresis before, after treatment, and after one month of follow up.

A statistical significant improvement in frequency of NE in both groups being more in group A but there is no statistically significant difference was detected between the two groups. A significant relapse rate after one month of follow in both groups but there is no statistically significant difference was detected between the two groups. Also, there was a statistical significant difference regarding improvement of frequency of NE more with patients with positive surgical history of tonsillectomy in both groups.

This study concluded that both Posterior tibial nerve stimulation and Desmopressin are viable treatment options in patients with primary mono-symptomatic nocturnal enuresis. PTNS is a good option if Desmopressin is contraindicated, fear of it's side effects or ineffective. We should tailor the treatment according to the child and caregiver's condition. Relapse in some responders in both groups with time suggests the need for maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

Aged between 5 and 13 years old .

* Experiencing more than two wetting episodes per week .
* Normal urinalysis results .
* Unremarkable urinary tract ultrasaound .
* Normal physical examination.

Exclusion Criteria:

* Diurnal enuresis .

  * Faecal soiling .
  * Cardiovascular disease .
  * Renal disorder .
  * Neurological disorders .
  * Urinary tract infection

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Posterior tibial nerve stimulation Vs desmopressin In children with primary monosymptomatic Nocturnal enuresis | 4 months
  Comparative study to show the effect of posterior tibial nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Hany A Morsi, Professor, Study Director — Cairo University
Locations (1):
- Abo ElRish children hospital, Cairo, Egypt